CLINICAL TRIAL: NCT03748888
Title: Physical Exercise, Cardiovascular Adaptation Monitoring in Pregnancy
Brief Title: Physical Exercise Cardiovascular Adaptation Monitoring in Pregnancy (PE-CAMP Study)
Acronym: PE-CAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Olga Roldan-Reoyo, Principal Investigator, Swansea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 663830-SU-079; 17/WA/0414 (Other: REC Reference)
Record Dates: First submitted 2018-11-13; First posted 2018-11-21 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Pregnancy Related; Pregnant Women; Maternal-Fetal Relations
Keywords: Cardiovascular system; Antenatal physical activity; Maternal heart rate; Foetal heart rate

STUDY DESIGN:
Intervention Model Description: The present study will involve two study groups.
  1. Exercise group (EG). Pregnant women allocated in the EG will receive and intervention based on a supervised antenatal physical activity programme during 20-24 weeks. They must be enrolled in the study between their 12-16 weeks of gestation.
  2. Control group (CG). Pregnant women allocated in CG will not receive any intervention. They will maintain standard health care during pregnancy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): An antenatal physical activity (APA) programme will be designed for participants in the exercise group.
  Interventions: Behavioral: Exercise group
- Control Group (No Intervention): Sedentary participants.

INTERVENTIONS:
Behavioral: Exercise group — An antenatal physical activity (APA) programme will be designed for participants in the exercise group.
  The APA will last for 20-24 weeks. Participants in the EG must enrol in the APA between their 12-16 weeks of gestation.
  The APA programme has a frequency of three times a week, which involves aerobic, strength and stretching exercises. The intensity of the APA programme is individually calculated for each participant based on their pre-pregnancy fitness level. Single sessions of the APA programme last 50-60min.
  Arms: Exercise group

SUMMARY:
The main theme of this study focuses on providing evidence of the impact of antenatal physical activity on maternal/foetal cardiovascular changes during pregnancy and maternal cardiovascular adaptations during the early postpartum period.

DETAILED DESCRIPTION:
Overwhelming research supports the general benefit of antenatal physical activity (APA) for pregnant women, but there is a lack of knowledge about the influence of exercise on cardiovascular physiology in healthy and overweight pregnant women and their foetuses. Also some research supports the theory of foetal programming; which establish that maternal habits during pregnancy will impact in-utero environment, so if this maternal habits are healthy ones they could improve foetal health.

Cardio vascular disease (CVD) was the top cause of death all over the world in 2015. In Wales CVD as cause of death is still one of the top ones. However, these statistics could be improved if people adopt healthier lifestyle habits, since 54% and 45% of Welsh women are overweight/obese or sedentary respectively. Pregnancy seems to be a teachable moment for women and the starting point of adopting healthy life-style habits. Therefore, by introducing Welsh pregnant women to exercise, there is the potential to improve their health and of their foetuses an also exert an exponential impact on future generations.

The main theme of this study focuses on providing evidence of the impact of APA on maternal/foetal cardiovascular changes during pregnancy and maternal cardiovascular adaptations during the early postpartum period.

This is a 3-year study carried out in Swansea University, Singleton Hospital.

The project leading to this application has received funding from the European Union's Horizon 2020 research and innovation programme under the Marie Sklodowska-Curie grant agreement No 663830.

Healthy pregnant women with no contraindications for exercise will be eligible for the study and those who want to participate in the project will be allocated into an exercise group (EG) or a control group (CG). EG participants will receive an intervention based on an APA during 20-24weeks, CG participants will follow their standard health care during pregnancy.

All participants must attend three cardiovascular assessment protocols (18-22 weeks & 32-36weeks during pregnancy, 12weeks postpartum). These protocols will involve maternal/foetal electrocardiograph and echocardiograph evaluation, heart-rate monitoring and moderate physical exercise (walking).

ELIGIBILITY:
Inclusion Criteria:

1. Women with healthy pregnancy
2. Aged 18-40 years
3. Single pregnancy
4. Pregnancy stage <= 16 weeks' gestation at the point of consent.
5. Two or fewer previous term pregnancies (as physiology can be altered by multiple pregnancies).

Exclusion Criteria:

1. Known complications of pregnancy
2. Known contraindications for physical exercise
3. Known major cardiovascular or respiratory pathology
4. Three or more previous term pregnancies
5. Inability to communicate in English or Welsh.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in maternal cardiac output during and after pregnancy. | 18 and 36 weeks of gestation, 12 weeks postpartum.
  Maternal cardiac output at rest, during exercise and after exercise measured in L/min would be recorded from study participants to analyse and compare potential changes inter and intra group.
Changes in maternal heart rate during and after pregnancy. | 18 and 36 weeks of gestation, 12 weeks postpartum.
  Maternal heart rate at rest and after exercise would be recorded in beats per minute to be analysed and compared inter and intra group.
Changes in maternal heart rate variability during and after pregnancy | 18 and 36 weeks of gestation, 12 weeks postpartum.
  Maternal heart rate variability at rest, during and after exercise would be measured by r to r interval. It would be recorded and analysed to compare inter and intra group changes.
Foetal heart rate | 36 weeks pregnancy
  Foetal heart rate baseline would be measured at rest, during and after exercise. It would be analysed and compared in between groups.

SECONDARY OUTCOMES:
Changes in active pregnant women energy expenditure | 18 and 36 weeks pregnancy.
  Data obtained from accelerometer devices worn by exercise group participants.
Changes in sedentary pregnant women energy expenditure | 18 and 36 weeks pregnancy.
  Data obtained from accelerometer devices worn by control group participants.
Energy expenditure during the early postpartum period. | 12 weeks postpartum.
  Data obtained from accelerometer devices worn by all participants in the study.
Gestational weight gain. | 36 weeks pregnancy.
  Weight gain during pregnancy measured in kilograms would be recorded to be compared in between study groups.
Changes in maternal body fat percentage during pregnancy. | 18 and 36 weeks pregnancy.
  Body fat percentage calculated from skinfold-thickness measures would be compared in between study groups.
Birth weight | Second week after birth.
  Birth weight from new borns recorded in kilograms would be collected from maternal records. It would be analysed and compared between groups.
Results from Qol-Grav questionnaire during second and third trimester of pregnancy. | 18 and 36 weeks pregnancy.
  The Qol-Grav questionnaire is a validated questionnaire used to measure quality of life in pregnant women. This questionnaire would be filled in by study participants and analysed to record their quality of life during the current pregnancy. Scores derived from the questionnaire would be analysed and compared between groups.
  The following total score scale is presented:
  9-18: Excellent quality of life. 19-27: Very good quality of life. 28-36: Good quality of life. 37-45: Not very good quality of life.
Pre-pregnancy physical activity levels recorded by the modified physical activity questionnaire. | 12 weeks pregnancy.
  Participants' pre-pregnancy physical activity levels would be registered using the modified physical activity questionnaire. This questionnaire records information about activities performed for the three months before pregnancy. Intensity of the activity would be recorded using three different levels of intensity (low, moderate and vigorous). Average time spent in each activity would be recorded in minutes. These values would be used to measure time and intensity spent in physical activity before pregnancy, and would be compared between groups.
Pregnancy physical activity levels during first trimester recorded by the modified physical activity questionnaire. | 12 weeks pregnancy.
  Participants' physical activity levels during the first trimester of pregnancy would be registered using the modified physical activity questionnaire. This questionnaire records information about activities performed during the first three months of pregnancy. Intensity of the activity would be recorded using three different levels of intensity (low, moderate and vigorous). Average time spent in each activity would be recorded in minutes. These values would be used to measure time and intensity spent in physical activity during pregnancy, and would be compared between groups.
Pregnancy physical activity levels during second and third trimester recorded by the modified physical activity questionnaire. | 36 weeks pregnancy.
  Participants' physical activity levels during the second and third trimester of pregnancy would be registered using the modified physical activity questionnaire. This questionnaire records information about activities performed during the second an third trimesters of pregnancy. Intensity of the activity would be recorded using three different levels of intensity (low, moderate and vigorous). Average time spent in each activity would be recorded in minutes. These values would be used to measure time and intensity spent in physical activity during pregnancy, and would be compared between groups.
Changes in quality of sleep during pregnancy. | 18 and 36 weeks of pregnancy.
  Two questionnaires would be used to measure participants' quality of sleep during their pregnancy. These questionnaires are the Pittsburgh Sleep Quality Index and the Insomnia Severity Index.
Quality of sleep during postpartum. | 12 weeks postpartum.
  Two questionnaires would be used to measure participants' quality of sleep during the postpartum period. These questionnaires are the Pittsburgh Sleep Quality Index and the Insomnia Severity Index.
Sleep patterns in the three months old infant | 12 weeks postpartum.
  The Brief Screening Questionnaire for Infant Sleep Problems would be used to register sleep patterns in the three months old infants born from study participants. Items recorded in the questionnaire are the following: sleep arrangement, time spent sleeping during the day and night, number of wakings per night, mode of falling asleep, time spent in wakefulness and normal time of falling asleep at night.

OTHER OUTCOMES:
Type of birth. | 2 weeks postpartum.
  Type of delivery such as vaginal, cesarean section or instrumental birth would be recorded from maternal records after birth.
Type of analgesia used during labour | 2 weeks postpartum.
  Type of analgesia (pharmacological or non-pharmacological) used during labour would be recorded from maternal records after birth.
New born's Apgar score | 2 weeks postpartum.
  Apgar score is a scale that measures health in the new born. This scale focuses on five parameters (skin colour, heart rate, reflexes and responsivness, muscular tone, and breathing rate), each of them rated from 0 to 2. This test is performed at the first and fifth minute of new born's life. Scores above 7 are consider normal, scores below 7 indicates that the new born needs medical attention. Scores from both tests (1min and 5min) would be recorded from maternal records after birth.
Changes in maternal hand grip strength during pregnancy. | 18 and 36 weeks of pregnancy.
  Maternal hand grip strength would be measured using a hand grip dynamometer. This test would be performed during the second and third trimester of pregnancy.
Maternal hand grip strength during postpartum. | 12 weeks postpartum.
  Maternal hand grip strength would be measured using a hand grip dynamometer. This test would be performed during the postpartum period.
Changes in maternal upper body range of motion during pregnancy. | 18 and 36 weeks of pregnancy.
  Maternal upper body flexibility during second and third trimester would be measured using the back scratch test. This test measures how close the hands can be brought together behind the back.
Maternal upper body range of motion during postpartum. | 12 weeks postpartum.
  Maternal upper body flexibility during the early postpartum would be measured using the back scratch test. This test measures how close the hands can be brought together behind the back.

CONTACTS AND LOCATIONS:
Overall Officials: MICHAEL J LEWIS, Prof, Study Chair — Swansea University
Locations (1):
- Singleton Hospital, Maternity Unit, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carpenter RE, Emery SJ, Uzun O, Rassi D, Lewis MJ. Influence of physical exercise on baroreceptor sensitivity during pregnancy. J Matern Fetal Neonatal Med. 2017 Mar;30(5):514-519. doi: 10.1080/14767058.2016.1179275. Epub 2016 May 12. PMID 27098455
- [Result] Carpenter RE, D'Silva LA, Emery SJ, Uzun O, Rassi D, Lewis MJ. Changes in heart rate variability and QT variability during the first trimester of pregnancy. Physiol Meas. 2015 Mar;36(3):531-45. doi: 10.1088/0967-3334/36/3/531. Epub 2015 Feb 18. PMID 25690105